CLINICAL TRIAL: NCT00861406
Title: An Exploratory Study of Adjuvant Therapy of Pegylated Interferon-Alfa 2b Plus Melanoma Peptide Vaccine in Patients With Resected Stage II and III (N1a, N2a) Melanoma
Brief Title: Adjuvant Therapy of Pegylated Interferon- 2b Plus Melanoma Peptide Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006-0816; NCI-2012-01652 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2009-03-12; First posted 2009-03-13 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-02

CONDITIONS: Melanoma
Keywords: Melanoma; Stage II melanoma; Pegylated Interferon-alfa 2b; PEG Interferon alfa-2b; PEG Intron; Melanoma Peptide Vaccine; GP100 Vaccine; gp100; peptide vaccine; Leukapheresis; Immune-cell response
MeSH Terms: conditions — Melanoma | interventions — peginterferon alfa-2b

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental): Pegylated Interferon alfa-2b (Once week x 4 weeks) + GP-100 Peptide
  Interventions: Drug: Pegylated Interferon-Alfa 2b (PEG Intron); Drug: GP-100 Peptide Vaccine
- Group 2 (Experimental): Pegylated Interferon alfa-2b (Once week x 8 weeks) + GP-100 Peptide
  Interventions: Drug: Pegylated Interferon-Alfa 2b (PEG Intron); Drug: GP-100 Peptide Vaccine
- Group 3 (Experimental): Pegylated Interferon alfa-2b (Once week x 12 weeks) + GP-100 Peptide
  Interventions: Drug: Pegylated Interferon-Alfa 2b (PEG Intron); Drug: GP-100 Peptide Vaccine

INTERVENTIONS:
Drug: Pegylated Interferon-Alfa 2b (PEG Intron) — Group 1:
  6 mcg/kg by injection under skin once weekly for 4 weeks, followed by Maintenance Phase of 3 mcg/kg weekly for 20 weeks.
  Group 2:
  6 mcg/kg by injection under skin once weekly for 8 weeks, followed by Maintenance Phase of 3 mcg/kg weekly for 16 weeks.
  Group 3:
  6 mcg/kg by injection under skin once weekly for 12 weeks followed by Maintenance Phase of 3 mcg/kg weekly for 12 weeks.
  Other Names: Peginterferon alfa-2b
Drug: GP-100 Peptide Vaccine — Injection under skin once every 3 weeks (Weeks 1, 4, 7, 10, 13, 16, 19, and 22), for a total of 8 injections.
  Other Names: melanoma peptide gp100 vaccine

SUMMARY:
The goal of this clinical research study is to find the best dosing schedule of a combined treatment of PEG Intron® (pegylated Interferon-alfa 2b) plus a peptide vaccine (gp100) that may help improve immune response in patients that had Stage II or Stage III melanoma and are free of the disease. The safety and tolerability of this drug combination will also be studied. Researchers also want to collect long-term follow-up information.

DETAILED DESCRIPTION:
The Study Drugs:

Pegylated Interferon alfa-2b is a protein made by the human immune system that helps to fight viral infections and regulate cell function.

Gp100 is a protein that is found on melanoma cells. In laboratory studies, the gp100 vaccine has been shown to stimulate the immune system to "recognize" and kill melanoma cells that have gp100 on their cell surfaces.

Evaluation of Immune cell response to vaccine:

Blood (about 3-1/2 tablespoons) will be drawn on Weeks 4, 7,10,13,16,19, and 22 for tests to check the response of your immune system to the vaccine, before each injection. These tests are for research purposes only and will not be used to make decisions about your medical care.

Parts of the Study:

There are 2 parts to this study, an Induction Phase and a Maintenance Phase. The Induction Phase treatment is the first course of treatment used to stimulate ("turn on") an immune-cell response to fight cancer and to learn the body's response to the treatment. The Maintenance Phase treatment is continued therapy and is used to maintain the immune-cell response and to help keep the disease in remission.

Study Groups:

If participant is found to be eligible to take part in this study, they will be randomly assigned (as in the roll of dice) to 1 of 3 treatment groups. Participant will have an equal chance of being assigned to one of each of the groups. Participants in each group will receive the same dose levels of pegylated Interferon alfa-2b and gp100. The difference between each group will be the dosing schedule of pegylated Interferon alfa-2b.

Every week, participant will give themselves the pegylated Interferon alfa-2b either in the clinic or at home, and the gp100 will be given to participant every 3 weeks by the research nurse in the clinic. Participant will be shown how to give yourself Pegylated Interferon alfa-2b at home.

Pegylated Interferon alfa-2b will be given immediately after the GP-100 Peptide Vaccine injection.

Participants in Group 1 will take pegylated Interferon alfa-2b at a certain dose level once a week for 4 weeks (in the Induction Phase), followed by once a week for 20 weeks in the Maintenance Phase (when the drug will be taken at a lower dose level than during Induction).

Participants in Group 2 will take pegylated Interferon alfa-2b at a certain dose level once a week for 8 weeks (in the Induction Phase), followed by once a week for 16 weeks in the Maintenance Phase (when the drug will be taken at a lower dose level than during Induction).

Participants in Group 3 will take pegylated Interferon alfa-2b at a certain dose level once a week for 12 weeks (in the Induction Phase), followed by once a week for 12 weeks in the Maintenance Phase (when the drug will be taken at a lower dose level than during Induction).

Study Treatment:

Participant will take pegylated Interferon alfa-2b as an injection just under their skin. Participant will receive gp100 as an injection just under their skin once every 3 weeks.

On Week 1, PEG-Intron will be given right after GP-100 Peptide Vaccine injection in the clinic. Participant will be observed for at least 30 minutes after both GP-100 Peptide Vaccine and PEG-Intron Injections.

On Weeks 4, 7, 10, 13, 16, 19, and 22 (+/- 1 day, not counting institutional holidays), GP-100 peptide will be given in the clinic. Participant will be observed for at least 30 minutes after GP-100 Peptide Vaccine injection. Participant should give the PEG-Intron to themselves within 24 hours of GP-100 Peptide Vaccine injection. The injection of gp100 will be given in two separate areas of participant's limbs, such as in an upper arm or thigh. It will be given in the same area each time.

Length of Study:

Participant will remain on this study for up to 25 weeks, unless the disease comes out of remission or they experience intolerable side effects.

End-of-Treatment Visit:

At the end of study treatment (approximately 3 weeks after the last injection of gp100), participant will have the following tests:

* Participant will have a review of their general health and any medical problems they may be having.
* Participant will have a physical exam, including measurement of their vital signs.
* Blood (about 1 tablespoon) will be drawn for routine tests.
* Participant will have the leukapheresis repeated.
* Participant will have a CT scan of chest, stomach, and pelvis, and they will have an MRI or CT scan of the brain.

While participant is on this study no steroids will be allowed while on treatment.

This is an investigational study. Pegylated Interferon alfa-2b is FDA approved and commercially available for the treatment of chronic hepatitis C. Gp100 is not FDA approved or commercially available. At this time, the combination use of pegylated Interferon alfa-2b plus gp100 is being used for research purposes only in this study.

Up to 30 participants will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be free of disease after surgical resection for American Joint Committee on Cancer (AJCC) stage II or III (N1a) melanoma (T2b, T3a, T3b, T4a, T4b and N1a or N2a). Diagnosis must be confirmed by the Pathology Department of MD Anderson Cancer Center.
2. Patients must be HLA-A0201 positive.
3. Patients must be fully recovered from surgery, for at least one month, but not more than 90 days after surgery and before study entry.
4. Patients must have no other malignancies. Patients with prior history of any in situ cancer, lobular carcinoma of the breast in situ, cervical cancer in situ, atypical melanocytic hyperplasia or Clark I melanoma in situ or basal or squamous skin cancer are eligible. Patients with other malignancies are eligible, if they have been continuously disease-free for 5 years prior to the time of study entry.
5. Patients must be >/= 18 years of age.
6. Patients must give signed written informed consent.
7. Women of childbearing potential (WOCBP) must not be pregnant (negative urine human chorionic gonadotropin (HCG) within 2 weeks of treatment) or lactating. A WOCBP has not undergone a hysterectomy or who has not been naturally postmenopausal for at least 24 consecutive months (i.e., who has had menses at any time in the preceding 24 consecutive months).
8. Women of childbearing potential and sexually active males must be counseled to use an accepted and effective method of contraception (including abstinence) while on treatment and for a period of 3 months after completing or discontinuing treatment. Simultaneous use of two contraceptive methods such as, intrauterine device (IUD) or condom and contraceptive jelly is considered the accepted method of contraception.
9. Patients must have Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
10. Patients must have white blood cell count (WBC) >/= 3,000/mm3, platelet count >/= 100,000/mm3, and hemoglobin >/= 9 g/dL or 5.6 mmole/L obtained within 2 weeks of study entry.
11. Patients must have AST, ALT, LDH, alkaline phosphatase, and bilirubin within institutional upper limit (IUL) of normal and serum creatinine < 2.0 mg/dl or < 140 micromol/L all obtained within 2 weeks of study entry. Patients with Gilbert's Disease may have bilirubin </= to 2 x (ULN).
12. Patients must have a CT of chest, abdomen, pelvis, and a MRI or CT scan of the brain performed within 4 weeks of study entry.

Exclusion Criteria:

1. Patients with clinical, radiological/laboratory or pathological evidence of incompletely resected melanoma or any distant metastatic disease.
2. Patients with autoimmune disorders or receiving immunosuppressive therapy including chemotherapy, steroids or methotrexate.
3. Patients requiring consistent use of antihistamines or non-steroidal anti-inflammatory drugs.
4. Patients with a history of active ischemic heart disease or cerebro-vascular disease, congestive heart failure (NYHA class >2) or anginal syndrome requiring ongoing medical treatment.
5. Patients have a diagnosis or evidence of organic brain syndrome or significant impairment of basal cognitive function or any psychiatric disorder that might preclude participation in the protocol. Any questionable patients will be reviewed by the investigator or attending physician.
6. Patients having prior radiotherapy, chemotherapy or any immunotherapy including, tumor vaccines, interferon, interleukins, levamisole or other biologic response modifiers for any type of cancer.
7. Patients with a history of central nervous system (CNS) demyelinating, inflammatory disease or hereditary or acquired grade 2 or higher peripheral neuropathy.
8. Patients with any other significant medical or surgical condition or psychiatric disorder, which includes any serious psychiatric illness that has not been adequately controlled despite intervention (with our without medication) with known history of HIV or hepatitis infection may interfere with the completion of this trial or with the evaluation of safety and efficacy of the study compound.
9. Patients with thyroid dysfunction not responsive to therapy.
10. Patients with pre-existing psychiatric condition including, but not limited to: a. History of severe depression, including the following: 1) Hospitalization for depression 2) Electroconvulsive therapy for depression 3) Depression that resulted in a prolonged absence from work and/or significant disruption of daily functions. b. Suicidal or homicidal ideation and/or suicidal or homicidal attempt. c. History of severe psychiatric disorders (eg. psychosis, post-traumatic stress disorder or mania). d. Past history or current use of lithium and/or antipsychotic drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2009-03-10 (Actual); Primary Completion 2017-02-24 (Actual); Study Completion 2017-02-24 (Actual)

PRIMARY OUTCOMES:
Patient Maximum T-cell Levels During 24-Week Treatment | Patient's T-cell levels assessed every 3 weeks using a tetramer assay.

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Jen Hwu, MD, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org